CLINICAL TRIAL: NCT03458130
Title: A Phase 2, Randomized, Placebo-controlled, Dose-ranging Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AG10 in Patients With Symptomatic Transthyretin Amyloid Cardiomyopathy
Brief Title: Study of AG10 in Amyloid Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eidos Therapeutics, a BridgeBio company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG10-201
Record Dates: First submitted 2018-02-07; First posted 2018-03-08 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Familial ATTR-CM (ATTRm-CM, or FAC); Wild-type ATTR-CM (ATTRwt-CM)

STUDY DESIGN:
Intervention Model Description: A randomized, doubleblind, placebo-controlled, dose-ranging design is considered to be the most appropriate study design for meeting this objective. On the basis of information gained from previous clinical experience with AG10, the doses used in this study will be selected to determine the dose with the better safety and tolerability profile.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AG10 Low Dose (Active Comparator): AG10 400mg tablets twice daily for 28 days
  Interventions: Drug: AG10
- AG10 High Dose (Active Comparator): AG10 800mg tablets twice daily for 28 days
  Interventions: Drug: AG10
- Placebo (Placebo Comparator): Placebo tablets twice daily for 28 days
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: AG10 — TTR stabilizer
  Arms: AG10 High Dose; AG10 Low Dose
Drug: Placebo Oral Tablet — Nonactive control
  Arms: Placebo

SUMMARY:
This prospective, randomized, multicenter, double-blind, parallel group, placebo-controlled, dose-ranging study will evaluate the safety, tolerability, PK (Pharmacokinetic) and PD (Pharmacodynamic) of AG10 compared to placebo administered on a background of stable heart failure therapy. Screening and randomization will be followed by a 28-day blinded, placebo-controlled treatment period.

DETAILED DESCRIPTION:
A Phase 2, Randomized, Placebo-controlled, Dose-ranging Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AG10 in Patients with Symptomatic Transthyretin Amyloid Cardiomyopathy.

The primary objective of this study is to evaluate the safety and tolerability of AG10 administered to adult patients with symptomatic transthyretin amyloid cardiomyopathy (ATTRCM).

This study will be a Phase 2, randomized, placebo-controlled, dose-ranging study in 45 male and/or female patients with symptomatic ATTR-CM aged 18 through 90 years.

If all doses are well tolerated, the duration of each patient's participation in the study will be 28 days of treatment. In addition, there will be a 28-day screening period before treatment and a 30-day follow-up period before the final Follow-up Visit.

This prospective, randomized, multicenter, double-blind, parallel group, placebo-controlled, dose-ranging study will evaluate the safety, tolerability, PK and PD of AG10 compared to placebo administered on a background of stable heart failure therapy. Screening and randomization will be followed by a 28-day blinded, placebo-controlled treatment period. secondary objectives of this study are: to characterize the pharmacokinetics (PK) of AG10 administered orally twice daily in patients with symptomatic ATTRCM, and to describe the pharmacodynamic (PD) properties of AG10 as assessed by established assays of transthyretin (TTR) stabilization, including Fluorescent Probe Exclusion (FPE) assay and Western blot, and to describe the Pharmacokinetic Pharmacodynamic (PKPD) relationship of AG10 in adult patients with symptomatic ATTRCM.

Eligible patients will be randomized in a 1:1:1 ratio to placebo or one of two different doses of AG10 administered twice daily. A minimum of 30% of patients enrolled will be mutant ATTR-CM.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
2. Be a male or female ≥18 to ≤90 years of age.
3. Have an established diagnosis of ATTR-CM with either wild-type transthyretin or a variant transthyretin genotype (assessed by genotyping, with patients with concurrent monoclonal gammopathy of undetermined significance requiring a confirmatory test using mass spectrometry) as defined by either positive endomyocardial biopsy or positive technetium pyrophosphate scan.
4. Have a history of heart failure evidenced by at least one prior hospitalization for heart failure or clinical evidence of heart failure (without hospitalization) requiring medical management.
5. Have New York Heart Association (NYHA) Class II-III symptoms.
6. Male patients and female patients of childbearing potential who engage in heterosexual intercourse must agree to use appropriate method(s) of contraception.
7. For patients taking cardiovascular medical therapy, with the exception of diuretic dosing, must be on stable doses (defined as no greater than 50% dose adjustment and no categorical changes of medications) for at least 2 weeks prior to Screening.

Exclusion Criteria:

1. Acute myocardial infarction, acute coronary syndrome or coronary revascularization within 90 days prior to Screening.
2. Experienced stroke within 90 days prior to Screening.
3. Has hemodynamic instability at Screening or Randomization that, in the judgment of the Principal Investigator (PI), would pose too great a risk for participation in the study.
4. Has estimated glomerular filtration rate (GFR) <30 mL/min/1.73 m2 at Screening.
5. Is likely to undergo heart transplantation within the next year.
6. Has confirmed diagnosis of light-chain amyloidosis.
7. Has abnormal liver function tests at Screening, defined as Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) >3 × upper limit of normal (ULN) or total bilirubin >2 × ULN.
8. Has abnormalities in clinical laboratory tests at Screening or Randomization that, in the judgment of the PI, would pose too great a risk for participation in the study.
9. Known hypersensitivity to study drug (AG10 or placebo), its metabolites, or formulation excipient
10. Current treatment with diflunisal, tafamidis, green tea, doxycycline, tauroursodeoxycholic acid (TUDCA)/Ursodiol, Patisiran or Inotersen within 14 days or 5 half-lives of the prior investigational agent (whichever is longer) prior to Screening.
11. Females who are pregnant or breastfeeding. Lactating females must agree to discontinue nursing before the study drug is administered. A negative serum pregnancy test at Screening and a negative urine pregnancy test at Randomization visit are required for female patients of childbearing potential.
12. In the judgment of the investigator, has any clinically significant ongoing medical condition that might jeopardize the patient's safety or interfere with the study, including participation in another investigational drug or investigational device study within the 30 days prior to Screening with potential residual effects that might confound the results of this study.
13. Has any laboratory abnormality or condition that, in the investigator's opinion, could adversely affect the safety of the patient or impair the assessment of study results.
14. Has any condition that, in the opinion of the investigator, would preclude compliance with the study protocol such as a history of substance abuse, alcoholism or a psychiatric condition.
15. Has participated in another investigational study within 14 days or 5 half-lives of the prior investigational agent (whichever is longer) prior to screening. Exceptions can be made in the case of observational and/or registry studies upon consultation with the Medical Monitor.
16. Current treatment with, or chronic use of, a proton pump inhibitor (PPI) or histamine-receptor 2 (H2) antagonist within 14 days or 5 half-lives of the prior agent (whichever is longer) prior to Screening.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-10-05 (Actual); Study Completion 2018-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MARK MCGOVERN, RN, Study Director — Eidos Therapeutics, a BridgeBio company
Locations (13):
- United States (13):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - Stanford University, Palo Alto, California
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Northwestern University, Chicago, Illinois
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Judge DP, Heitner SB, Falk RH, Maurer MS, Shah SJ, Witteles RM, Grogan M, Selby VN, Jacoby D, Hanna M, Nativi-Nicolau J, Patel J, Rao S, Sinha U, Turtle CW, Fox JC. Transthyretin Stabilization by AG10 in Symptomatic Transthyretin Amyloid Cardiomyopathy. J Am Coll Cardiol. 2019 Jul 23;74(3):285-295. doi: 10.1016/j.jacc.2019.03.012. Epub 2019 Mar 15. PMID 30885685

RESULTS

PARTICIPANT FLOW:
Groups:
- AG10 400mg: AG10 400mg twice daily for 28 days; tablets
  AG10: Transthyretin (TTR) stabilizer
- AG10 800mg: AG10 800mg twice daily for 28 days; tablets
  AG10: Transthyretin (TTR) stabilizer
- Placebo: Placebo twice daily for 28 days; tablets
Period: Overall Study
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Started | 16 | 16 | 17
Screening | 16 | 16 | 17
Double Blind Treatment | 16 | 16 | 17
Follow-Up | 16 | 16 | 17
Completed | 16 | 16 | 17
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AG10 400mg: AG10 400mg twice daily for 28 days; tablets
  AG10: TTR stabilizer
- AG10 800mg: AG10 800mg twice daily for 28 days; tablets
  AG10: TTR stabilizer
- Total: Total of all reporting groups
Arm/Group | AG10 400mg | AG10 800mg | Placebo | Total
Number analyzed (Participants) | 16 | 16 | 17 | 49
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.8 (5.65) | 75.4 (6.81) | 73.2 (7.35) | 74.1 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 0 | 4
  Male | 14 | 14 | 17 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 14 | 14 | 15 | 43
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race (NIH/OMB): American Indian or Alaska Native | 0 | 0 | 0 | 0
  Race (NIH/OMB): Asian | 1 | 0 | 0 | 1
  Race (NIH/OMB): Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
  Race (NIH/OMB): Black or African American | 4 | 3 | 3 | 10
  Race (NIH/OMB): White | 10 | 12 | 13 | 35
  Race (NIH/OMB): Other | 1 | 1 | 1 | 3
  Race (NIH/OMB): More than one race | 0 | 0 | 0 | 0
  Race (NIH/OMB): Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 17 | 49
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/meters squared] | 25.42 (3.284) | 26.29 (3.705) | 27.05 (3.604) | 26.27 (3.528)
Height [Mean (Standard Deviation); unit: Centimeters] | 172.68 (7.055) | 175.59 (9.738) | 174.52 (8.220) | 174.27 (8.317)
TTR Genotype Status [Count of Participants; unit: Participants] — Composition of the TTR gene
  Participants
    Wild Type | 10 | 11 | 14 | 35
    Mutant | 6 | 5 | 3 | 14
    Other | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: Kilograms] | 75.93 (12.080) | 81.71 (15.948) | 82.34 (12.018) | 80.04 (13.478)

OUTCOME MEASURES:

1. Primary Outcome: Change in Diastolic Blood Pressure
Description: Change in Diastolic Blood Pressure from Baseline to Day 28 (Postdose)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
mm Hg
  Change in Diastolic Blood Pressure from Baseline to Day 28 (Predose) | -3.1 (10.06) | -3.3 (11.19) | -4.3 (7.78)
  Change in Diastolic Blood Pressure from Baseline to Day 28 (Postdose) | -2.6 (9.66) | 0.3 (8.54) | -4.9 (9.17)

2. Primary Outcome: Change in Heart Rate
Description: Change in Heart Rate from Baseline to Day 28 (Postdose)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
beats/minute
  Change in heart rate from Baseline to Day 28 (Predose) | -2.7 (6.88) | -3.8 (6.55) | -0.4 (6.34)
  Change in heart rate from Baseline to Day 28 (Postdose) | -7.3 (9.84) | -4.9 (5.84) | -1.1 (8.89)

3. Primary Outcome: Change in Respiratory Rate
Description: Change in Respiratory Rate from Baseline to Day 28 (Postdose)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: breaths/minute
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
breaths/minute
  Change in Respiratory Rate from Baseline to Day 28 (Predose) | -0.1 (2.23) | -0.8 (3.12) | -0.4 (2.35)
  Change in Respiratory Rate from Baseline to Day 28 (Postdose) | -0.7 (1.68) | -1.1 (3.11) | -1.1 (2.93)

4. Primary Outcome: Change in Temperature
Description: Change in Temperature from Baseline to Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
degrees Celsius
  Change in Temperature from Baseline to Day 28 (Predose) | 0.17 (0.793) | 0.06 (0.316) | -0.08 (0.506)
  Change in Temperature from Baseline to Day 28 (Postdose) | 0.22 (0.781) | -0.02 (0.357) | 0.02 (0.194)

5. Primary Outcome: Change in Systolic Blood Pressure
Description: Change in Systolic Blood Pressure from Baseline to Day 28
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
mm Hg
  Change in Systolic Blood Pressure from Baseline to Day 28 (Predose) | -2.7 (12.05) | -8.1 (12.36) | -5.3 (13.50)
  Change in Systolic Blood Pressure from Baseline to Day 28 (Postdose) | -2.8 (18.41) | -4.1 (8.88) | -3.4 (17.51)

6. Secondary Outcome: Number of Participants With Threshold Levels of Overall % Stabilization >= 95% and >= 99% by Fluorescent Probe Exclusion (FPE)
Description: In specialized lab tests on patient samples that measure the stability of the healthy form of TTR, both doses of AG10 were able to reach near complete stabilization.
Time Frame: Day 1 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | AG10 400mg | AG10 800mg | Placebo
Number analyzed (Participants) | 16 | 16 | 17
Participants
  % Stabilization > = 95 % | 14 | 15 | 0
  % Stabilization > = 99 % | 11 | 13 | 0

7. Secondary Outcome: Pharmacokinetic (PK): Steady State Trough Concentration of AG10
Description: Non-fluctuating minimal amount of AG10 in blood at Day 14 and Day 28
Time Frame: Day 14 and Day 28
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AG10 400mg | AG10 800mg
Number analyzed (Participants) | 16 | 16
ng/mL
  AG10: PK Plasma Concentration at Day 14 (Pre-Dose) | 1924.4 (837.3) | 2257.3 (982.81)
  AG10: PK Plasma Concentration at Day 28 (Pre-Dose) | 1841.3 (483.88) | 2439.4 (900.08)

ADVERSE EVENTS:
Time Frame: Onset date on or after first dose of study drug and not more than 30 days after last dose of study drug, up to day 58.
Arm/Group | AG10 400mg | AG10 800mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 2/17
Other Adverse Events (participants affected / at risk) | 10/16 | 11/16 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG10 400mg (N=16) | AG10 800mg (N=16) | Placebo (N=17)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AG10 400mg (N=16) | AG10 800mg (N=16) | Placebo (N=17)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 1 (2) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 2 (2)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2)
Fluid Retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3)
Fluid Overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema Peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Venous Pressure Jugular Increased (Investigations) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the results by the PI will be subject to mutual agreement between the PI and the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT03458130/Prot_001.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/30/NCT03458130/SAP_002.pdf